CLINICAL TRIAL: NCT02037529
Title: A Randomized Phase III Trial of Eribulin Compared to Standard Weekly Paclitaxel as First- or Second-Line Therapy for Locally Recurrent or Metastatic Breast Cancer
Brief Title: Eribulin Mesylate or Paclitaxel as First- or Second-Line Therapy in Treating Patients With Recurrent Stage IIIC-IV Breast Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Total enrollment number is being lowered
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU011201I; NCI-2016-02048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU011201I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2023-09-06 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-08

CONDITIONS: Breast Adenocarcinoma; HER2/Neu Negative; Invasive Breast Carcinoma; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (eribulin mesylate) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm B (paclitaxel) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
  Arms: Arm A (eribulin mesylate)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well eribulin mesylate or paclitaxel work as first- or second-line therapy in treating patients with stage IIIC-IV breast cancer that has come back. Drugs used in chemotherapy, such as eribulin mesylate and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that patient-reported Patient-Report Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) data will be able to detect differences in symptoms between participants treated witheribulin mesylate (eribulin) and standard weekly paclitaxel at 12 weeks.

II. To validate rs7349683 in EPHA5 as a predictor of peripheral neuropathy from treatment with a microtubule targeting agent (i.e., eribulin or paclitaxel).

SECONDARY OBJECTIVES:

I. To compare overall survival, progression free survival (PFS), objective response rate (ORR), duration of response (DOR), and time to treatment failure (TTF) in patients receiving eribulin versus standard weekly paclitaxel.

II. To compare the 12 month rate of disease progression in patients receiving eribulin versus standard weekly paclitaxel.

III. To evaluate the clinical value and feasibility of collecting patient-reported symptom toxicity information via the Patient-Report Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).

IV. To further validate the PRO-CTCAE sensory neuropathy items. V. To compare patient reported neurotoxicity between arms using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Chemotherapy-Induced Peripheral Neuropathy 20 (CIPN20) instrument.

VI. To assess the toxicities in patients receiving eribulin versus standard weekly paclitaxel.

CORRELATIVE OBJECTIVES:

I. To compare new metastasis free survival in patients receiving eribulin versus standard weekly paclitaxel.

II. To explore the relationship between common single nucleotide polymorphisms in FGD4, FZD3, and VAC14 as predictors of peripheral neuropathy from treatment with a microtubule targeting agent (i.e., eribulin or paclitaxel).

III. To evaluate circulating nucleosomes and the apoptosis associated M30 neo-epitope as potential biomarkers associated with clinical benefit from treatment with eribulin specifically or the microtubule dynamics inhibitors in general.

VI. To evaluate tubulin isotype expression, mutations, and signaling pathway modifications in tumor tissue as potential biomarkers associated with clinical benefit from treatment with eribulin specifically or the microtubule dynamics inhibitors in general.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent document signed and dated by patient
* Histologic confirmation of invasive adenocarcinoma originating in the breast
* Stage IV disease or stage IIIC disease (using the 7th edition American Joint Committee on Cancer [AJCC] criteria) not amenable to local therapy
* Clinical or radiographic evidence of disease progression
* Documentation of HER2 negative breast cancer at the time of protocol registration; (Note: HER2 negativity is defined as 0 or 1+ by immunohistochemistry OR nonamplified or equivocal by fluorescence in situ hybridization [FISH]; status may be defined on the basis of historic results on the breast primary or a metastatic site, whichever is most recent; repeat biopsies are not required for participation in this protocol)
* Known hormone receptor status at the time of protocol registration; (Note: estrogen receptor [ER] and/or progesterone receptor [PgR] status are considered positive with a cut-off of >= 1% invasive tumor cells; status may be defined on the basis of historic results on the breast primary or a metastatic site, whichever is most recent; repeat biopsies are not required for participation in this protocol)
* Patients must demonstrate resolution of all toxicities related to prior chemotherapy, endocrine therapy, targeted therapy, or biologic therapy to grade =< 1, including peripheral neuropathy, with the exception of alopecia (any grade permissible)
* No more than one prior chemotherapy regimen for advanced or metastatic breast cancer is allowed; prior chemotherapy for metastatic disease must have been completed >= 14 days prior to randomization

  * Any single agent therapy, and any combination of cytotoxic, endocrine, biological targeted agents, and/or humanized antibodies, scheduled to be administered as a preplanned treatment, given concomitantly, sequentially or both, is considered one regimen
  * Planned neoadjuvant chemotherapy and postoperative adjuvant chemotherapy is considered one regimen
  * If the dosing of one or more of the chemotherapy components of a regimen must be reduced for toxicity, the modified version of the original regimen is not considered a new regimen
  * If one or more of the chemotherapy components of a regimen must be omitted for toxicity, the modified version of the original regimen is not considered a new regimen
  * If one of the chemotherapy components of a regimen must be replaced with another similar drug of the same therapeutic class, the modified version of the original regimen is not considered a new regimen; however, if a new component, dissimilar to any of the original components, is added to the regimen, the modified version is considered a new regimen
  * If chemotherapy is interrupted for surgery or radiotherapy and then continues with an unchanged schedule and components, treatment is considered as one regimen despite the interruption
* Prior treatment may include a taxane as per the following criteria:

  * Prior taxane (including paclitaxel) in the adjuvant or neoadjuvant setting is allowed, provided that the interval between the completion of (neo)adjuvant therapy and disease recurrence is > 12 months
  * Prior taxane in the metastatic setting is allowed, provided that the agent administered in the metastatic setting was not standard paclitaxel
* Any number of prior endocrine therapies is allowed and must be discontinued prior to randomization
* Any number of biologic therapies (e.g., bevacizumab) or immunotherapies is allowed in the absence of co-administered chemotherapy and must have been completed >= 28 days prior to randomization
* Prior treatment with an investigational agent is allowed but must have been completed >= 28 days prior to randomization with resolution of all treatment-related toxicities to grade =< 1.
* Minor surgical procedures must be completed >= 7 days prior to randomization with documentation of adequate recovery from associated complications to grade =< 1; these include (but are not limited to) laparoscopy, thoracoscopy, bronchoscopy, mediastinoscopy, endoscopic ultrasonography, skin biopsy, percutaneous needle biopsy, and routine dental procedures; as a precautionary measure, it is recommended, but not strictly required, that placement of a central venous access device, thoracentesis, or paracentesis be done 7 days before the initiation of protocol directed chemotherapy with documentation of adequate recovery from associated complications to grade =< 1
* Major surgical procedures and open biopsies must be completed >= 28 days prior to randomization with documentation of adequate recovery from associated complications to grade =< 1
* Prior radiotherapy must be completed >= 14 days prior to randomization with documentation of adequate recovery from associated toxicities to grade =< 1
* Treatment with bisphosphonates or denosumab is allowed and recommended per the standard of care
* Therapeutic anticoagulation is allowed for patients on a stable dose of warfarin or low molecular weight heparin
* Measurable disease is defined as at least one lesion that can be accurately measured with the longest diameter as >= 1.0 cm by computed tomography (CT) scan or >= 1.0 cm with calipers by clinical examination; the exceptions to these criteria are pathologic lymph nodes, which must be >= 1.5 cm in the short axis when assessed by CT scans with slice thickness =< 0.5 cm
* Non-measurable lesions include the following: small lesions (longest diameter < 1.0 cm for all lesions other than pathologic lymph nodes, which are >= 1.0 cm and < 1.5 cm in the short axis), bone metastases, pleural effusions, pericardial effusions, ascites, inflammatory breast disease, leptomeningeal disease, lymphangitis pulmonis, lymphangitis cutis, and abdominal masses not followed by CT or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of > 12 weeks
* Patients with a history of resected brain metastases are eligible only if they are asymptomatic and have stable MRI scans for 3 consecutive months, including =< 28 days of study registration
* Patients who receive stereotactic radiosurgery or whole brain radiation for brain metastases are eligible only if they are asymptomatic and have stable MRI scans for 3 consecutive months, including =< 28 days of study registration
* Obtained =< 7 days prior to registration: Absolute neutrophil count >= 1500/uL
* Obtained =< 7 days prior to registration: Platelet count >= 100,000/uL
* Obtained =< 7 days prior to registration: Hemoglobin >= 9 g/dL
* Obtained =< 7 days prior to registration: Total bilirubin =< 1.5 times the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert?s syndrome
* Obtained =< 7 days prior to registration: Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferases [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN except in the case of liver metastases, where =< 5 x ULN is allowed
* Obtained =< 7 days prior to registration: Creatinine =< 2.0 mg/dL or creatinine clearance > 50 mL/min
* Obtained =< 7 days prior to registration: Corrected QT (QTc) interval =< 500 msec on the baseline electrocardiogram
* Negative pregnancy test done =< 72 hours prior to registration for women of childbearing potential only; Note: all female subjects will be considered to be of child-bearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically (i.e., bilateral tubal ligation >= 1 menstrual cycle prior to randomization, or have undergone a hysterectomy and/or bilateral oophorectomy)

  * Female subjects of child-bearing potential must agree to use highly effective contraception during the study treatment and for 3 months after the final dose of study treatment; female subjects exempt from this requirement are subjects who practice total abstinence; if currently abstinent, the subject must agree to use a double barrier method of contraception (i.e., condom and occlusive cap [diaphragm or cervical/vault caps]) with spermicide or until they are established on highly effective contraception for at least one menstrual cycle if they become sexually active during the study treatment and for 3 months after the final dose of study treatment
  * Highly effective contraception includes:

    * Placement of intrauterine device or system
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) with spermicide
    * Vasectomized partner with confirmed azoospermia
  * Male subjects and their female partner who are of child-bearing potential (as defined above), and are not practicing total abstinence, must agree to use highly effective contraception during study treatment and for 3 months after the final dose of study treatment; if currently abstinent, the subject must agree to use a double barrier method of contraception if they become sexually active, or until they are established on highly effective contraception as described above
* Ability to complete questionnaire(s) independently or with assistance
* Willingness to provide blood and tissue samples for correlative research purposes; (Note: these tissue samples are from archived tissue, if available; new biopsies are not required)
* Ability to comprehend and respond to questions using a telephone keypad

Exclusion Criteria:

* Prior malignancy, other than carcinoma in situ of the cervix and non-melanoma skin cancers, unless the prior malignancy was diagnosed and definitively treated >= 5 years previously, there is no subsequent evidence of recurrence, and the patient is considered by a physician to be at < 30% risk of relapse
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Presence of a serious nonhealing wound, ulcer, or bone fracture
* History of Common Terminology Criteria for Adverse Events (CTCAE) grade >= 3 hypersensitivity to paclitaxel or Cremophor EL
* Pre-existing peripheral neuropathy grade ?= 2 at registration
* Significant cardiovascular impairment (e.g., New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia)
* Subjects with known positive human immunodeficiency virus (HIV) status
* History of stroke or transient ischemic attack =< 6 months prior to registration
* History of uncontrolled seizures; (Note: patients are eligible for the study if the seizures are well controlled with standard medications)
* Severe or uncontrolled intercurrent illness/infection
* Concurrent administration of any other investigational agent considered to have potential efficacy in the treatment of breast cancer
* Prior exposure to eribulin mesylate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2024-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Minetta C Liu, Principal Investigator — Academic and Community Cancer Research United
Locations (39):
- United States (39):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner NCI Community Oncology Research Program, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Essentia Health NCI Community Oncology Research Program, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Heartland Cancer Research CCOP, St Louis, Missouri
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Mission Hospital-Saint Joseph Campus, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Women and Infants Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Eribulin): Patients receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Started | 101 | 100
Completed | 100 | 96
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel) | Total
Number analyzed (Participants) | 101 | 100 | 201
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [53 to 70] | 62 [53.5 to 68] | 62 [53 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 100 | 199
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 95 | 95 | 190
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 20 | 32
  White | 85 | 76 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dose Level Triggering a Grade 2 or Higher Neuropathy Event.
Description: To validate rs7349683 in EPHA5 as a predictor of peripheral neuropathy from treatment with a microtubule targeting agent (i.e., eribulin or paclitaxel) over the first 6 months of treatment we will compare the median cumulative dose level triggering a grade 2 or higher neuropathy event.
Time Frame: 6 months
Population: All treated patients
Measure: Median (Inter-Quartile Range); unit: mg/m^2
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 100 | 98
mg/m^2 | 39.25 [33.2 to 75.6] | 3950 [2442 to 6186]

2. Primary Outcome: Mean Change in Patient Reported PRO-CTCAE
Description: To demonstrate that patient-reported PRO-CTCAE data will be able to detect differences in symptoms between participants treated with eribulin and standard weekly paclitaxel at 12 weeks we will compare the mean change of overall Pro-CTCAE score by treatment arm. The overall Pro-CTCAE score is a normalized score scaled from 20 questions, each with a possible 1-5 patient selection, creating an overall score (0-100) where 0 represents the best outcome and 100 represents the worst possible outcome. The mean change from baseline to week 12 is reported.
Time Frame: 12 weeks
Population: Treated patients that completed baseline and week 12 patient reported PRO-CTCAE packets.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 98 | 92
score on a scale | 3.72 (0.57) | 3.77 (0.61)

3. Secondary Outcome: Overall Survival (OS)
Description: The primary analysis will use the stratified log-rank tests, as described for overall survival. As a secondary analysis we will use a multivariable Cox proportional hazard model to estimate adjusted hazard ratios for eribulin mesylate over standard weekly paclitaxel, study stratification factors, and covariates for known prognostic factors, including disease free interval and visceral versus non-visceral metastases. Survival functions will be summarized using the Kaplan-Meier method according to treatment group.
Time Frame: 81 months
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
months | 18.1 [15.4 to 22.1] | 16.4 [14.5 to 23.3]
Statistical Analysis 1: Comparison: Arm A (Eribulin) vs Arm B (Paclitaxel); Test type: Superiority; p = 0.5623, Log Rank

4. Secondary Outcome: Objective Tumor Response Rate
Description: Objective tumor response rate is assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Time Frame: 64 months
Population: All treated patients
Measure: Number; unit: proportion of participants
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 100 | 98
proportion of participants | 0.14 | 0.21

5. Secondary Outcome: Duration of Response
Description: Will be summarized using the Kaplan-Meier method. Will use a two-sided type I alpha of 0.05, and point estimates will be reported with 95% confidence intervals. Duration of response is the time between a tumor response and progression.
Time Frame: 75 months
Population: All patients that achieved a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 29 | 32
Months | 13.7 [9.0 to 19.6] | 14.1 [8.4 to 19.8]

6. Secondary Outcome: Time to Treatment Failure
Description: Will use a two-sided type I alpha of 0.05, and point estimates will be reported with 95% confidence intervals.
Time Frame: 64 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
Months | 5.3 [3.7 to 5.6] | 4.9 [3.2 to 5.5]

7. Secondary Outcome: Incidence of Treatment Related Adverse Events
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). Events determined to be possibly or probably attributed to a medical treatment suggest there is evidence to indicate a causal relationship between the drug and the adverse event. The number of patients that experienced an AE, of any grade, determined to be possibly or probably attributed to a medical treatment will be reported by arm.
Time Frame: 64 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
Participants | 94 | 90

8. Secondary Outcome: Time to New Metastasis
Description: Will be summarized using the Kaplan-Meier method. Will use a two-sided type I alpha of 0.05, and point estimates will be reported with 95% confidence intervals.
Time Frame: 81 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
Months | 8.2 [5.7 to 16.9] | 8.7 [6.0 to 11.3]
Statistical Analysis 1: Comparison: Arm A (Eribulin) vs Arm B (Paclitaxel); Test type: Superiority; p = 0.9840, Log Rank

9. Secondary Outcome: Progression Free Survival Assessed by RECIST 1.1 Criteria
Description: Will be summarized using the Kaplan-Meier method. Will use a two-sided type I alpha of 0.05, and point estimates will be reported with 95% confidence intervals. Progression free survival time is the time from date of randomization to the date of first progression or death.
Time Frame: 80 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
Months | 5.7 [5.4 to 7.1] | 5.9 [5.3 to 8.3]
Statistical Analysis 1: Comparison: Arm A (Eribulin) vs Arm B (Paclitaxel); Test type: Superiority; p = 0.5968, Log Rank

10. Secondary Outcome: Patients With Reported Neurotoxicity
Description: Additional analyses will include the previously described analysis conducted over the first 24 weeks; a comparison of the incidence of patient-reported maximum score >= 3 between arms through 12 and 24 weeks using chi-squared testing for each item; and a comparison of the time to patient-reported score >= 3 between arms using Kaplan-Meier and log-rank analyses. Further, these three endpoints will be compared between patient- and clinician-report overall and within arms using appropriate paired analyses.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
Number analyzed (Participants) | 101 | 100
Participants | 26 | 31

11. Secondary Outcome: Validation of PRO-CTCAE Sensory Neuropathy Item
Description: The PRO-CTCAE sensory neuropathy items will be further validated by computing Pearson correlations between each item, severity and interference, and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Chemotherapy-Induced Peripheral Neuropathy 20 (CIPN20 )sensory scale score at baseline, 12 and 24 weeks.
Time Frame: At baseline, 12, and 24 weeks
Population: This analysis was pre-specified in the Statistical Analysis Plan to be conducted overall and not separately for each of the arms. Only patients that fully filled out and submitted their PRO-CTCAE and EORTC QLQ-CIPN20 packets are included in this analysis.
Measure: Number; unit: Pearson correlation
Groups:
- All Patients: The PRO-CTCAE sensory neuropathy items will be further validated by computing Pearson correlations between each item and the EORTC QLQ-CIPN20 sensory scale score at baseline, 12 and 24 weeks.
Arm/Group | All Patients
Number analyzed (Participants) | 154
Pearson correlation
  Baseline - Severity | 0.72
  Baseline - interference | 0.67
  Week 12 - severity: number analyzed (Participants) | 90
  Week 12 - severity | 0.71
  Week 12 - interference | 0.51
  Week 24 - severity: number analyzed (Participants) | 38
  Week 24 - severity | 0.79
  Week 24 - interference | 0.85

12. Other Pre Specified Outcome: New Metastasis Free Survival
Description: Will be summarized using the Kaplan-Meier method according to treatment group.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 64 months and mortality was followed for 81 months.
Arm/Group | Arm A (Eribulin) | Arm B (Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 80/101 | 79/100
Serious Adverse Events (participants affected / at risk) | 30/101 | 30/100
Other Adverse Events (participants affected / at risk) | 99/101 | 95/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Eribulin) (N=101) | Arm B (Paclitaxel) (N=100)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 3 (3) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Eribulin) (N=101) | Arm B (Paclitaxel) (N=100)
Anemia (Blood and lymphatic system disorders) | 32 (32) | 39 (39)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 5 (5) | 7 (7)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 4 (4)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 3 (3) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 13 (13)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 50 (50) | 40 (40)
Dental caries (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 33 (33) | 43 (43)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 9 (9)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 5 (5)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 21 (21) | 15 (15)
Nausea (Gastrointestinal disorders) | 45 (45) | 46 (46)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth discoloration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (19) | 20 (20)
Chills (General disorders) | 4 (4) | 2 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 13 (13) | 15 (15)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 70 (70) | 61 (61)
Fever (General disorders) | 7 (7) | 8 (8)
Flu like symptoms (General disorders) | 3 (3) | 5 (5)
Gait disturbance (General disorders) | 2 (2) | 3 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (3) | 3 (3)
Malaise (General disorders) | 1 (1) | 1 (1)
Neck edema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 7 (7)
Pain (General disorders) | 33 (33) | 25 (25)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2) | 3 (3)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Breast infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3) | 10 (10)
Lung infection (Infections and infestations) | 3 (3) | 3 (3)
Mucosal infection (Infections and infestations) | 2 (2) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 2 (2)
Papulopustular rash (Infections and infestations) | 2 (2) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 6 (6)
Skin infection (Infections and infestations) | 7 (7) | 5 (5)
Upper respiratory infection (Infections and infestations) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 7 (7) | 7 (7)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 13 (13) | 12 (12)
Alkaline phosphatase increased (Investigations) | 12 (12) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 18 (18) | 13 (13)
Blood bilirubin increased (Investigations) | 3 (3) | 2 (2)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 5 (5)
ECG QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 11 (11) | 11 (11)
Neutrophil count decreased (Investigations) | 43 (43) | 22 (22)
Platelet count decreased (Investigations) | 11 (11) | 5 (5)
Weight gain (Investigations) | 2 (2) | 2 (2)
Weight loss (Investigations) | 14 (14) | 5 (5)
White blood cell decreased (Investigations) | 25 (25) | 18 (18)
Anorexia (Metabolism and nutrition disorders) | 40 (40) | 36 (36)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (13) | 10 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5) | 10 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 11 (11) | 10 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 15 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 16 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 20 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 2 (2)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 10 (10) | 12 (12)
Dysgeusia (Nervous system disorders) | 7 (7) | 8 (8)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 21 (21)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 6 (6)
Movements involuntary (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 5 (5) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (2) | 2 (2)
Paresthesia (Nervous system disorders) | 5 (5) | 7 (7)
Peripheral motor neuropathy (Nervous system disorders) | 4 (4) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 48 (48) | 50 (50)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 12 (12) | 12 (12)
Confusion (Psychiatric disorders) | 3 (3) | 4 (4)
Depression (Psychiatric disorders) | 9 (9) | 13 (13)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 34 (34) | 40 (40)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 5 (5)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 25 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 31 (31)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 62 (62) | 62 (62)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 4 (4)
Hot flashes (Vascular disorders) | 11 (11) | 11 (11)
Hypertension (Vascular disorders) | 9 (9) | 14 (14)
Hypotension (Vascular disorders) | 5 (5) | 4 (4)
Lymphedema (Vascular disorders) | 4 (4) | 8 (8)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT02037529/Prot_SAP_000.pdf